CLINICAL TRIAL: NCT03745703
Title: MOCHA Moving Forward: a CBPR Investigation of Chronic Disease Prevention in Older, Low-income African-American Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: University of Massachusetts, Worcester (Other); YMCA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-4898
Record Dates: First submitted 2018-11-09; First posted 2018-11-19 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2021-11

CONDITIONS: Chronic Disease of Cardiovascular System; Multiple Chronic Conditions; Chronic Disease
MeSH Terms: conditions — Multiple Chronic Conditions; Chronic Disease

STUDY DESIGN:
Intervention Model Description: The study design uses a wait-list control to test the effectiveness and relative effectiveness of a community-driven MOCHA intervention, including discussions of salient health topics (such as stress and anger management) and an enhanced version MOCHA+, which incorporates narrative communication strategies to strenghten comprehnsion, retention and motivation.
Who Masked: Participant
Masking Description: Participants are randomly assigned to either the MOCHA standard arm or to the enhanced MOCHA+ arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MOCHA (Experimental): Behavioral: 12-week trial with 3 sessions per week with one small group discussion session of critical issues affecting African-American men's health each week combined with two aerobic exercise sessions each week
  Interventions: Behavioral: MOCHA
- MOCHA+, "Stories Matter" (Experimental): Behavioral: 12-week trial with 3 sessions per week with one small group discussion session of critical issues affecting African-American men's health each week combined with two aerobic exercise sessions each week
  Interventions: Behavioral: MOCHA
- Wait-list control (No Intervention): There is no intervention to be administered during the 12-week wait-list control period

INTERVENTIONS:
Behavioral: MOCHA — (see above)
  Other Names: MOCHA+
  Arms: MOCHA; MOCHA+, "Stories Matter"

SUMMARY:
The overall goal of the research is to discover how to reduce chronic disease health disparities among older (ages 35-70) low-income African-American men more effectively. To achieve this goal, the investigators are conducting formative exploratory research with middle-aged, low-income African-American men; testing two versions of a novel community-developed intervention, MOCHA and MOCHA+ (where MOCHA+ is a modified version of the "standard" MOCHA program, modified to incorporate narrative communication strategies); and advancing the development of a Minority Stress Model through statistical modelling to test the relative contributions of hypothesized explanatory variables identified in the formative research phase of the project.

DETAILED DESCRIPTION:
Low-income, African-American men continue to be disproportionately burdened by chronic diseases and associated morbidities and mortalities. Primary modifiable and interrelated causes of chronic disease include high levels of stress, low levels of physical activity, and malnutrition. There are few demonstrated effective, preventive interventions that are culturally relevant and gender appropriate for low-income, African-American men.

Local community concerns about health disparities led to a year-long series of community-wide discussions and planning that resulted in the creation of Men of Color Health Awareness (MOCHA) project. Started in 2010, in an unusual public-private partnership between the YMCA and the state Department of Public Health, MOCHA's mission is to improve the health and wellbeing of men of color in Springfield, MA and surrounding areas. MOCHA runs a 12-week program with 15-20 men per cohort to decrease chronic disease vulnerability and bolster resilience among low-income, African-American men, by addressing exercise, eating habits, and stress stemming from impoverished economic conditions, racial and class discrimination, and gender role strain. The MOCHA Steering Committee contacted a group of health disparities researchers at the University of Massachusetts School of Public Health and Health Sciences in 2012, requesting assistance in documenting the impact of MOCHA on the community.

Over 350 men ages 40-60 years have completed the MOCHA program and preliminary data indicate that the program has decreased weight, body fat percentage, and systolic blood pressure; increased self-reported fitness and vitality scores; and decreased mean stress scores on the Cohen Perceived Stress scale by 19%. Based on these preliminary data, the research team proposes to rigorously test MOCHA program effectiveness and to identify the causal pathways through which it impacts outcomes.

In addition, the MOCHA Steering Committee has expressed strong interest in strengthening the quality of their program, by incorporating narrative strategies for communicating key health concepts and information into the existing program. Current research of the investigators provides strong evidence that culture-centered narrative strategies are more effective in producing positive health effects than didactic presentations. The collaborating partners have pilot tested the feasibility of developing digital stories with the MOCHA Steering Committee, and with this proposal, the investigators are mutually excited about the possibility of integrating narrative communication strategies into the MOCHA program, henceforth called MOCHA+.

To test the effectiveness of the existing MOCHA chronic disease prevention program in decreasing stress and compare its effectiveness with a new to-be-developed MOCHA+ program (that integrates narrative communication strategies), the research team proposes to conduct a randomized-controlled trial with three arms: MOCHA, MOCHA + and wait-list control comparison groups. Using a community-based participatory research approach, the three specific aims of the proposed research are thus to:

1. Further refine a Minority Stress Model developed by Co-PI Graham, to capture and explain the dynamic, reciprocal and synergistic interactions of factors affecting the health of low-income African-American men;
2. (a) Determine the effectiveness of the MOCHA program in decreasing stress among low-income African-American men, as measured by both self-report (Cohen's Perceived Stress Scale) and bio-physiological measures of cortisol (assessed in hair samples); and (b) Determine whether the MOCHA+ program is significantly more effective than the MOCHA program in decreasing stress among low-income African-American men, on these same measures;
3. Assess the effects of the MOCHA and MOCHA+ interventions on mediating variables along hypothesized causal pathways identified through intervention mapping and the construction of a logic model, based on the Minority Stress Model finalized in achieving Aim 1.

The proposed research will proceed in two stages. During the first 18 months, phase one of the study will focus on (a) formative research designed to further elaborate the minority stress model and (b) the incorporation of narrative communications strategies into the MOCHA+ intervention. In phase two, the investigators will recruit 240 low-income African-American men between 35-65 years of age over a three-year period to participate in a randomized controlled trial, with three arms: MOCHA, MOCHA+, or wait-list control. The primary research endpoint is bio-physiological assessment of the ELISA cortisol hair-test (average hormone levels over the past 3 months), administered at pre, post, and 3 month follow-up, as well as self-reported stress levels using Cohen's Perceived Stress scale. Secondary outcomes include the bio-physiological indicators of blood pressure and BMI.

The proposed research will determine the effectiveness of MOCHA in reducing stress and whether it can be further strengthened by introducing narrative communication strategies. The results of the proposed research will contribute to the development of an enhanced theoretical model of factors affecting low-income African-American male health and to the evidence base of effective interventions aimed at chronic disease prevention and control programs in this population.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet all of the inclusion criteria in order to be eligible to participate in the study.

Inclusion criteria include:

1. self-identification as black, African-American, or bi-racial including black man;
2. age between 35-70 years;
3. insufficient or low income;
4. lived in Springfield area for the previous 6 months;
5. Informed consent;
6. Understand study procedures; and
7. Ability to comply with study procedures for the entire length of the study

Exclusion Criteria:

Exclusion criteria include:

1. BMI>40;
2. BP>179/ 119;
3. PTSD scale score >50
4. Physical or movement l imitations wherein unable to perform 60 minutes of moderately vigorous physical activity 2 times per week

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 261 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Stress, as measured by Cohen's Perceived Stress Scale | Six months
  Subjective measure of stress is being collected to evaluate the impact of the MOCHA intervention
Stress, as measured by cortisol levels in fingernail samples | Six months
  Objective measure of stress is being collected to evaluate the impact of the MOCHA intervention

SECONDARY OUTCOMES:
High blood pressure | Six months
  High blood pressure
Body Mass Index | Six months
  Weight and height will be combined to report BMI in kg/m.

CONTACTS AND LOCATIONS:
Overall Officials: David Buchanan, DrPH, Principal Investigator — UMass School of Public Health & Health Sciences
Locations (2):
- United States (2):
  - University of Massachusetts, Amherst, Massachusetts
  - City of Springfield, Springfield, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graham LF, Scott L, Lopeyok E, Douglas H, Gubrium A, Buchanan D. Outreach Strategies to Recruit Low-Income African American Men to Participate in Health Promotion Programs and Research: Lessons From the Men of Color Health Awareness (MOCHA) Project. Am J Mens Health. 2018 Sep;12(5):1307-1316. doi: 10.1177/1557988318768602. Epub 2018 Apr 26. PMID 29695204
- [Background] Valdez LA, Gubrium AC, Markham J, Scott L, Hubert A, Meyer J, Buchanan D. A culturally and gender responsive stress and chronic disease prevention intervention for low/no-income African American men: The MOCHA moving forward randomized control trial protocol. Contemp Clin Trials. 2021 Feb;101:106240. doi: 10.1016/j.cct.2020.106240. Epub 2020 Dec 7. PMID 33301990